CLINICAL TRIAL: NCT03175679
Title: A Study of Adoptive Invariant Nature Killer T Cell Therapy for Relapsed/Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Adoptive Transfer of iNKT Cells for Treating Patients With Relapsed/Advanced HCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing YouAn Hospital (Other)
Responsible Party: Principal Investigator, LU JUN, Director of Hepatology and Cancer Biotherapy Ward, Beijing YouAn Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Beijing Youan Ethics[2017]05
Record Dates: First submitted 2017-05-24; First posted 2017-06-05 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Interleukin-2; Tegafur; gimeracil; potassium oxonate

STUDY DESIGN:
Intervention Model Description: Four planned loading dose of iNKT cells for 10 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- iNKT cell loading dose:3x10^7/m2 (Experimental): Autologous in vitro expanded iNKT cells in conjunction with IL-2 and along with lymphodepleting chemotherapy (Tegafur) will be administered to patients with advanced HCC.
  iNKT Cell Loading Dose：3x10^7/m2.
  IL-2: IL-2 will be given at a dose of 25,000 IU/kg/day for 5-14 days.
  Tegafur: Tegafur will be given at a dose of 40~60 mg bis in die (BID) 2 weeks.
  Interventions: Biological: iNKT cells; Drug: IL-2; Drug: Tegafur
- iNKT cell loading dose:6x10^7/m2 (Experimental): Autologous in vitro expanded iNKT cells in conjunction with IL-2 and along with lymphodepleting chemotherapy (Tegafur) will be administered to patients with advanced HCC.
  iNKT Cell Loading Dose：6x10^7/m2.
  IL-2: IL-2 will be given at a dose of 25,000 IU/kg/day for 5-14 days.
  Tegafur: Tegafur will be given at a dose of 40~60 mg bis in die (BID) 2 weeks.
  Interventions: Biological: iNKT cells; Drug: IL-2; Drug: Tegafur
- iNKT cell loading dose:9x10^7/m2 (Experimental): Autologous in vitro expanded iNKT cells in conjunction with IL-2 and along with lymphodepleting chemotherapy (Tegafur) will be administered to patients with advanced HCC.
  iNKT Cell Loading Dose：9x10^7/m2.
  IL-2: IL-2 will be given at a dose of 25,000 IU/kg/day for 5-14 days.
  Tegafur: Tegafur will be given at a dose of 40~60 mg bis in die (BID) 2 weeks.
  Interventions: Biological: iNKT cells; Drug: IL-2; Drug: Tegafur
- iNKT cell loading dose:1x10^10/m2 (Experimental): Autologous in vitro expanded iNKT cells in conjunction with IL-2 and along with lymphodepleting chemotherapy (Tegafur) will be administered to patients with advanced HCC.
  iNKT Cell Loading Dose：1x10^10/m2.
  IL-2: IL-2 will be given at a dose of 25,000 IU/kg/day for 5-14 days.
  Tegafur: Tegafur will be given at a dose of 40~60 mg bis in die (BID) 2 weeks.
  Interventions: Biological: iNKT cells; Drug: IL-2; Drug: Tegafur

INTERVENTIONS:
Biological: iNKT cells — The patients received different doses of in vitro-expanded autologous iNKT cells through intravenous infusion. The dosage was escalated from 3x10^7 cells/m2 to 6x10^7 cells/m2 to 9x10^7 cells/m2. The maximum tolerated dose (MTD) was defined as the last dose level, and the dosage would be up to 1x10^10 cells/m2 if no MTD was observed after a 3+3 design.
Drug: IL-2 — IL-2 will be given at a dose of 25,000 IU/kg/day for 5-14 days.
  Other Names: Human recombinated Interleukin-2
Drug: Tegafur — Tegafur will be given at a dose of 40~60 mg bis in die (BID) 2 weeks.
  Other Names: Gimeracil and Oteracil Potassium Capsules

SUMMARY:
This study enrolls patients who have relapsed/advanced hepatocellular carcinoma (HCC, BCLC stage C). The HCC tumor relapsed or metastasized through the body after standard treatment or the patients cannot receive standard treatment under current conditions. This research study uses special immune system cells called iNKT cells, a new experimental treatment.

The purpose of this study is to find the biggest dose of iNKT cells that is safe and tolerance, to see how long they last in the body, to learn the immunoresponse in the body, to learn the side effects are and to see if the iNKT cells will help people with relapsed/advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
PBMCs of enrolled patients were collected and then further separated by density gradient centrifugation. After washing three times, the cells were resuspended in serum-free medium with recombinant human IL-2 and α-GalCer. Restimulation with α-GalCer-pulsed autologous DCs was done on days 7. After 14 days of cultivation, the iNKT cells were harvested, washed thrice, and then resuspended in saline. The frequency of iNKT cells before and after cultured in vitro were determined by flow cytometry analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Patients with hepatocellular carcinoma (BCLC, stage C) proved by histopathology or proved by CT or MRI imaging system, relapsed after previous therapy and no effective therapies known at this time.
* Life expectancy of ≥ 12 weeks.
* WBC>3.5×10^9/L, LYMPH> 0.8×10^9/L, Hb>85g/L, PLT>50×10^9/L, Cre<1.5×the upper limit of normal value.
* iNKT>10/mL in peripheral blood mononuclear cell (PBMC).
* Able to understand and sign the informed consent.

Exclusion Criteria:

* Any uncontrolled systematic disease: hypertension, heart disease, and et al.;
* Portal vein tumor thrombus, central nervous system tumor metastasis, or combined with other tumors;
* Receiving radiochemotherapy, local therapy, or targeting drugs within 4 weeks prior to this treatment;
* Unstable immune systematic diseases or infectious diseases;
* Combined with AIDS or syphilis;
* Patients with history of stem cell or organ transplantation;
* Patients with allergic history to related drugs and immunotherapy;
* Patients with complications associated with liver diseases: moderate or severe pleural effusion, pericardial effusion, ascites, or gastrointestinal hemorrhage;
* Pregnant or lactating subjects;
* Unsuitable subjects considered by clinicians.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Lu, Director, Study Chair — Beijing YouAn Hospital
Locations (1):
- Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients diagnosed of HCC in the stage of BCLC B or C. But they don't have severe dysfunction of liver, kidney, heart and lung. Expected survival is more than 12weeks.
Pre-assignment Details: A total of 10 patients were recruited in this study from April 2017 to May 2018. Patient 1-8 received cell transfusion in stages according to the plan of 10%，30%，60% of them were used per infusion every other day, and patient 9 and 10 infused all of the cells at one-time.
Period: Overall Study
Arm/Group | iNKT Cell Loading Dose:3x10^7/m2 | iNKT Cell Loading Dose:6x10^7/m2 | iNKT Cell Loading Dose:9x10^7/m2 | iNKT Cell Loading Dose:1x10^10/m2.
Started | 3 | 3 | 3 | 1
Completed | 3 | 3 | 3 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 10 patients were enrolled in the experiment from April 2017 to May 2018.
Groups:
- iNKT Cell Loading Dose:1x10^10/m2: Autologous in vitro expanded iNKT cells in conjunction with IL-2 and along with lymphodepleting chemotherapy (Tegafur) will be administered to patients with advanced HCC.
  iNKT Cell Loading Dose：1x10^10/m^2 Cells.
  IL-2: IL-2 will be given at a dose of 25,000 IU/kg/day for 5-14 days.
  Tegafur: Tegafur will be given at a dose of 40~60 mg bis in die (BID) 2 weeks.
- Total: Total of all reporting groups
Arm/Group | iNKT Cell Loading Dose:3x10^7/m2 | iNKT Cell Loading Dose:6x10^7/m2 | iNKT Cell Loading Dose:9x10^7/m2 | iNKT Cell Loading Dose:1x10^10/m2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 10
Age, Categorical [Count of Participants; unit: Participants] — All enrolled patients take a physical examination before the study begins. And they are clearly diagnosed of hepatocellular carcinoma and in the stage of Barcelona Clinic Liver Cancer (BCLC) stage B/C. But they don't have severe dysfunction of liver, kidney, heart and lung. The diagnosis of hepatocellular carcinoma (BCLC stage B/C) was confirmed by CT, MRI. Expected survival is more than 12weeks.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 3 | 3 | 3 | 1 | 10
    >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 50 [50 to 60] | 51 [45 to 59] | 52 [37 to 59] | 53 [53 to 53] | 51.5 [37 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 1
  Male | 3 | 3 | 2 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 3 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
BCLC (Barcelona Clinic Liver Cancer ) stage [Count of Participants; unit: Participants] — All enrolled patients take a physical examination before the study begins. And they are clearly diagnosed of hepatocellular carcinoma and in the stage of Barcelona Clinic Liver Cancer (BCLC) stage B/C. The diagnosis of hepatocellular carcinoma (BCLC stage B/C) was confirmed by CT, MRI.
  Participants
    BCLC stage B | 0 | 0 | 1 | 1 | 2
    BCLC stage C | 3 | 3 | 2 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Defined as signs/symptoms, laboratory toxicities, and clinical events that are possibly, likely, or definitely related to study treatment Adverse events assessed according to NCI-CTCAE v4.0 criteria 2.
Time Frame: During the first 12 weeks, participants were assessed for adverse events every 2-4 weeks after infusion; after the first 12 weeks, participants were assessed for adverse events every 3 months, up to 20 months.
Population: Adverse events defined as the occurrence of toxicity events within 4 weeks after iNKT cells infusion. The severity of adverse events were divided into 5 levels.
Measure: Number; unit: events
Groups:
- iNKT Cell Loading Dose:3x10^7/m2: Autologous in vitro expanded iNKT cells in conjunction with IL-2 and along with lymphodepleting chemotherapy (Tegafur) will be administered to patients with advanced HCC.
  Autologous in vitro expanded iNKT cells in conjunction with IL-2 and along with lymphodepleting chemotherapy (Tegafur) will be administered to patients with advanced HCC.
  iNKT Cell Loading Dose：3x10^7/m2.
  IL-2: IL-2 will be given at a dose of 25,000 IU/kg/day for 5-14 days.
  Tegafur: Tegafur will be given at a dose of 40~60 mg bis in die (BID) 2 weeks.
Arm/Group | iNKT Cell Loading Dose:3x10^7/m2 | iNKT Cell Loading Dose:6x10^7/m2 | iNKT Cell Loading Dose:9x10^7/m2 | iNKT Cell Loading Dose:1x10^10/m2
Number analyzed (Participants) | 3 | 3 | 3 | 1
events
  Grade 1 | 12 | 2 | 8 | 4
  Grade 2 | 0 | 1 | 1 | 1
  Grade 3 | 2 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 1 | 1 | 2 | 1

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is the time that passes from the date that patient enrolled in the clinical trial and the date on which HCC progresses or the date on which the patient dies. HCC progression was evaluated by imaging according to the irRC standard. Progression is defined as a ≥25% increase in the nadir of the sum of target lesions.
Time Frame: Through study completion, an average of 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | iNKT Cell Loading Dose:3x10^7/m2 | iNKT Cell Loading Dose:6x10^7/m2 | iNKT Cell Loading Dose:9x10^7/m2 | iNKT Cell Loading Dose:1x10^10/m2
Number analyzed (Participants) | 3 | 3 | 3 | 1
Participants
  <6months | 1 | 1 | 2 | 0
  6-12months | 1 | 2 | 1 | 1
  >12months | 1 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Stabilized (SD) or Progressive (PD) Disease.
Description: Disease stabilization (SD) or progressive diseasee (PD) were valuated by imaging according to the irRC standard. Complete response (CR): Disappearance of all lesions; Partial response (PR): ≥50% decrease from baseline; SD: Neither CR or PD is met; PD≥25% increase in the nadir of the sum of target lesions.
Time Frame: 4 weeks, 8 weeks, 12 weeks and 24 weeks after cell infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | iNKT Cell Loading Dose:3x10^7/m2 | iNKT Cell Loading Dose:6x10^7/m2 | iNKT Cell Loading Dose:9x10^7/m2 | iNKT Cell Loading Dose:1x10^10/m2
Number analyzed (Participants) | 3 | 3 | 3 | 1
Participants
  At 4th week after cell infusion: SD | 3 | 3 | 3 | 1
  At 4th week after cell infusion: PD | 0 | 0 | 0 | 0
  At 8th week after cell infusion: SD | 2 | 3 | 1 | 1
  At 8th week after cell infusion: PD | 1 | 0 | 2 | 0
  At 12th week after cell infusion: SD | 2 | 3 | 1 | 1
  At 12th week after cell infusion: PD | 1 | 0 | 2 | 0
  At 24th week after: SD | 2 | 1 | 1 | 1
  At 24th week after: PD | 1 | 2 | 2 | 0

4. Secondary Outcome: Overall Survival (OS)
Description: OS is the time that passes from the date that patient enrolled in the clinical trial and the date on which the patient dies, according to the irRC standard.
Time Frame: Through study completion, up to 20 months.
Measure: Number; unit: participants
Arm/Group | iNKT Cell Loading Dose:3x10^7/m2 | iNKT Cell Loading Dose:6x10^7/m2 | iNKT Cell Loading Dose:9x10^7/m2 | iNKT Cell Loading Dose:1x10^10/m2.
Number analyzed (Participants) | 3 | 3 | 3 | 1
participants
  <6months | 1 | 0 | 2 | 0
  6-12months | 0 | 1 | 0 | 1
  >12months | 2 | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: During the first 12 weeks, participants were assessed for adverse events every 2-4 weeks after infusion; after the first 12 weeks, participants were assessed for adverse events every 3 months, up to 20 months.
Description: The severity of adverse events were divided into 5 levels according to the National Cancer Institute (NCI) Common Terminology Standard for Adverse Events (CTCAE) version 4.03.
Arm/Group | iNKT Cell Loading Dose:3x10^7/m2 | iNKT Cell Loading Dose:6x10^7/m2 | iNKT Cell Loading Dose:9x10^7/m2 | iNKT Cell Loading Dose:1x10^10/m2
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 2/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 2/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iNKT Cell Loading Dose:3x10^7/m2 (N=3) | iNKT Cell Loading Dose:6x10^7/m2 (N=3) | iNKT Cell Loading Dose:9x10^7/m2 (N=3) | iNKT Cell Loading Dose:1x10^10/m2 (N=1)
Cirrhosis and upper gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) — Not considered relatedto the iNKT cell therapy.
Refractory bile duct infection and toxic megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not considered relatedto the iNKT cell therapy.
Spontaneous rupture of the tumor (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not considered relatedto the iNKT cell therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iNKT Cell Loading Dose:3x10^7/m2 (N=3) | iNKT Cell Loading Dose:6x10^7/m2 (N=3) | iNKT Cell Loading Dose:9x10^7/m2 (N=3) | iNKT Cell Loading Dose:1x10^10/m2 (N=1)
Chills (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fever (Immune system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased platelet count (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Decreased neutrophil count (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased white blood cell count (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Increased blood bilirubin level (Hepatobiliary disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Increased alanine transaminase level (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Increased aspartate transaminase level (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Subcutaneous induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT03175679/Prot_SAP_000.pdf